CLINICAL TRIAL: NCT05820490
Title: ImpaCt Of Shiftwork on METabolic Flexibility and Skeletal Muscle Clocks
Acronym: COMET
Status: Recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1993997
Record Dates: First submitted 2023-02-28; First posted 2023-04-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Health
Keywords: metabolic flexibility; skeletal muscle circadian clock; fatty acid oxidation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We will sample muscle biopsies during the evening and morning time to examine diurnal shifts in skeletal muscle clock gene expression, which is a proxy of in vivo skeletal muscle circadian timing.
  We will also take serial blood draws every hour for 24 hours to assess changes in circulating hormones.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dayshift workers
  Interventions: Other: Whole Room Calorimeter; Other: Mixed-Meal Tolerance Test (MMTT); Other: Core Body Temperature; Other: Morningness-Eveningness Questionnaire; Procedure: Muscle Biopsy; Other: Serial Blood Sampling
- Nightshift workers
  Interventions: Other: Whole Room Calorimeter; Other: Mixed-Meal Tolerance Test (MMTT); Other: Core Body Temperature; Other: Morningness-Eveningness Questionnaire; Procedure: Muscle Biopsy; Other: Serial Blood Sampling

INTERVENTIONS:
Other: Whole Room Calorimeter — The indirect calorimetry system allows your oxygen / carbon dioxide exchange to be measured, thereby showing the number of calories burned.
Other: Mixed-Meal Tolerance Test (MMTT) — The MMTT is done to measure how much body handles a mixed meal.This test shake will raise blood sugar and cause the body to produce insulin.
Other: Core Body Temperature — Participants will be asked to swallow a core body temperature monitor prior to entering the whole room calorimeter. This monitor is used to record participants core body temperature.
Other: Morningness-Eveningness Questionnaire — Participants will fill out a questionnaire that asks about your preference for morning or evening.
Procedure: Muscle Biopsy — Participants will have two skeletal muscle biopsies (one in the evening and one in the morning). This procedure is used to sample muscle cells from the right and left leg Vastus Lateralis (thigh) muscle.
Other: Serial Blood Sampling — Participants will have blood sampled every hour for 24 hours to assess changes in circulating hormones.

SUMMARY:
The purpose of this study is to determine the impact of real-world shiftwork on metabolic flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45 yrs
* Employed as a healthcare worker in either dayshift (N=15) or nightshift work (N=30).
* Nightshift is defined as 12 months of consecutive nightshift work, who had 10 or more nightshifts per month (6 h between 10 PM and 8 AM, with no shift duration > 12 h).
* Dayshift is defined as 12 months of consecutive dayshift work, who had 10 or more dayshifts per month (6h between 8 AM and 10 PM, with no shift duration > 12 h).
* Weight Stable (+/- 3 kg over past 6 months)
* BMI between 18.5-29.9 kg/m2
* Understands the procedures and agrees to participate by giving written informed consent
* Willing and able to comply with scheduled visits, laboratory tests, and other study procedures including
* Only low to moderate caffeine users (<500 mg/day, or up to approximately 5 cups [1 cup=8 ounces] of coffee/day.

Exclusion criteria:

* Acute or chronic medical conditions or medication that would contraindicate participation in the research testing or could potentially affect metabolic function including, but not limited to:
* History or presence of cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, presence of cardiac pacemaker, implanted cardiac defibrillator)
* Type 1 or Type 2 diabetes mellitus
* Obesity (BMI ≥ 30 kg/m2)
* Bleeding and clotting disorders
* Uncontrolled hypertension (BP >160 mmHg systolic or >100 mmHg diastolic)
* Acute or chronic infections (such as TB, HIV, or Hepatitis)
* Renal insufficiency or nephritis (eGFR<60), nephritis, or chronic kidney disease
* Chronic obstructive pulmonary disease
* Thyroid dysfunction (suppressed TSH, elevated TSH <10 µIU/ml if symptomatic or elevated TSH >10 µIU/ml if asymptomatic)
* Liver disease (liver function tests > 2 x normal; including nonalcoholic steatohepatitis [NASH] and non-alcoholic fatty liver disease [NAFLD])
* Diagnosed or being treated for sleep disorders
* History of Cushing's disease or syndrome
* Pregnant or nursing females or females less than 6 months postpartum from the scheduled date of collection
* Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women) during screening
* Participation in studies involving investigational drug(s) within 30 days prior to Screening
* Gastrointestinal disorders (including inflammatory bowel disease or malabsorption, swallowing disorders, suspected or known strictures, fistulas or physiological/mechanical GI obstruction, history of gastrointestinal surgery, Crohn's disease or diverticulitis)
* Past or present history of psychiatric disease, including major depressive illness or bipolar disorder, as well as claustrophobia since part of the protocol will involve being confined to a small room for whole-body indirect calorimetry
* Unwilling or unable to eat foods provided in study procedures
* Nickel allergy
* Lidocaine allergy
* Any malignancy not considered cured, except basal cell carcinoma and squamous cell carcinoma of the skin (a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years)
* Use of antibiotics within 3 months of screening
* Illicit drug use (negative tests at screening)
* Regular smoking or regular nicotine use of any kind including chewing tobacco, snuff and vaping
* History of regular alcohol consumption exceeding 7 drinks/week for female participants or 14 drinks/week for male participants (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
* Excessive caffeine use (>500 mg/day, or exceeding 5 cups [1 cup= 8 ounces] of coffee/day)
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to Screening (participants may not donate blood any time during the study, through the final study day)
* Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study days.
* More than 1-day a week of intentional exercise

Excluded medications include, but are not limited to:

* Any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
* Medications that strongly impact bleeding, clotting, bruising, or platelets (e.g. blood thinner prescription medications)
* Recent change to medication and/or dosing in the past 3 months
* Chronic use of aspirin or other non-steroidal anti-inflammatory drugs, including COX-2 inhibitors

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will enroll normal weight and overweight, sedentary, but otherwise healthy adults employed in shiftwork.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Metabolic flexibility, or substrate switching capacity, will differ between dayshift and nightshift workers. | 30 days, including a two night stay
  Rates (change over time) of substrate oxidation will be assessed via whole-room indirect calorimetry during a 24h protocol that includes controlled meals and sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Erickson, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

REFERENCES:
- See also: AdventHealth Translational Research Institute website — https://www.adventhealthresearchinstitute.com/research/translational-research